CLINICAL TRIAL: NCT00820560
Title: A Phase I, Open-Label, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB007839 Following Multiple Oral Doses in Patients With Solid Tumors
Brief Title: Open-Label Study to Assess the Safety/Tolerability in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 7839-201
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors and Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INCB07839 100mg, immediate release (IR) capsules (Experimental)
  Interventions: Drug: INCB007839
- INCB07839 200 mg IR capsules (Experimental)
  Interventions: Drug: INCB007839

INTERVENTIONS:
Drug: INCB007839 — INCB007839 100 or 200 mg/dose as IR capsules

SUMMARY:
To establish the maximum tolerated dose (MTD) of INCB007839 given as multiple doses for 28 days and to determine if a higher MTD can be established when INCB007839 is administered in combination with prophylactic anticoagulation and with a 2 and a half day (5 doses) treatment interruption every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Either non-small cell lung cancer, hormone-refractory prostate cancer, colorectal cancer, breast cancer, or squamous cell cancer of the head and neck that is refractory to standard treatment or for which no effective treatment exists. The patient must have a life expectancy of 12 weeks or longer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Received any anticancer medications in the 28 days prior to receiving their first dose of study medication
* Evidence of venous thrombosis by flow Doppler examination at Screening
* A history of thrombosis or a coagulation disorder
* Patients with a contraindication to use of low dose warfarin and/or aspirin.
* Any unresolved toxicity greater than grade 2 from previous anticancer therapy, except for stable chronic toxicities not expected to resolve
* Brain metastases or spinal cord compression
* Impaired renal function
* Inadequate bone marrow reserve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Identify a maximum tolerable dose as measured through adverse event reporting, ECGs and laboratory assessments | Baseline through study completion

SECONDARY OUTCOMES:
Evaluation of response rates as measured by RECIST criteria | At Screening, Day 1 of all 28 day cycles beginning of each subsequent odd numbered cycle.
Evaluation of PSA laboratory values for response | Baseline and every visit through study termination
Evaluation of PD markers for HER2 and ErbB ligand levels | Measured at screening and Day 1 of all subsequent 28 days cycles and Day 15 of Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: William V Williams, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - Aurora, Colorado
  - Baltimore, Maryland
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee